CLINICAL TRIAL: NCT01604083
Title: European Transfusion Practice and Outcome Study A Multi-central Evaluation of Standard of Transfusion Care and Clinical Outcome for Elective Surgical Patients. Observational Study.
Brief Title: European Transfusion Practice and Outcome Study
Acronym: ETPOS
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: ETPOS
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2016-04

CONDITIONS: Surgery; Erythrocyte Transfusion; Habits; Anemia; Blood Coagulation Disorders
Keywords: transfusion; packed red blood cells (PRBC); Transfusion Practice; Transfusion habits; Outcome; elective surgery; ETPOS; ESA; European Society of Anaesthesiology
MeSH Terms: conditions — Habits; Anemia; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the ETPOS study is to describe differences in transfusion habits throughout Europe and to correlate these habits to perioperative outcome parameters. Special focus is put on the number of PRBCs (packed red blood cells) transfused and the ratio of PRBCs to other blood products or coagulation factors in the operating room. Furthermore the motivation of physicians to transfuse PRBC and blood products in the operating room will be investigated.

DETAILED DESCRIPTION:
In European patients undergoing elective non-cardiac surgery receiving at least one PRBC(packed red blood cells) during their surgery it is proposed to:

1. Evaluate evidence of differences in the standard of peri-operative transfusion care in different healthcare systems within Europe, and the use of blood conserving techniques.

   1. Evaluate the ratio of transfusion of PRBC to blood products in the operating room
   2. Evaluate which factors determine transfusion of PRBC (is it patient's haemodynamics / haemoglobin threshold/ pressure from the surgeon / acute brisk bleeding / else) and blood products (ratio to PRBC / POC (point of care) monitoring/ per protocol/ else) in the operating room
2. Evaluate whether there are factors in transfusion therapy that are associated with outcome (in-hospital mortality and unplanned admission to ICU(Intensive Care Unit).)

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing elective non-cardiac surgery commencing during the three-month period and who received at least one erythrocyte concentrate during their intra-operative stay.

Exclusion Criteria:

* Age < 18 years
* cardiothoracic surgery
* emergency trauma patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a non cardiothoracic, non emergency-trauma surgical procedure of participating hospital will be included, if they receive at least one pRBC. There are no further specific inclusion criteria. The only exclusion criteria will be age < 18 years and cardiothoracic and emergency trauma patients.
Sampling Method: Non-Probability Sample
Enrollment: 6066 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Amount of PRBC and blood products and coagulation factors transfused | The Time point at which outcome measure is assessed is during surgery at Day 0
  Amount of packed red blood cells and blood products and coagulation factors: fresh frozen plasmas (FFPs), platelets (PTs) and tranexamic acid transfused

SECONDARY OUTCOMES:
Factors determining transfusion of PRBC and blood products in different regions of Europe | The Time point at which outcome measure is assessed is during surgery at Day 0
  Reasons for transfusion of PRBC(packed red blood cells)and blood products in different regions of Europe
30-day mortality | The Time point at which outcome measure is assessed is at Day 30 after Surgery
  Assesses on Day 30 whether patient is still alive or has died between day zero (Surgery) day 30 after surgery
Unplanned admission to the ICU | The Time point at which outcome measure is assessed is at Day 30 after Surgery
  Assesses on day 30 whether the patient had a Unplanned admission to the Intensive care unit(ICU) following surgery (day 0) until the day 30
Type and frequency of usage of blood conserving techniques | The Time point at which outcome measure is assessed is at Day 0, on Surgery Day

CONTACTS AND LOCATIONS:
Overall Officials: Jens Meier, MD, Study Chair — General Hopsital Linz, Linz, Austria
Locations (9):
- University hospital "Merkur", Zagreb, Croatia
- Faculty Hospital Brno, Brno, Czechia
- North Estonian Center, Tallinn, Estonia
- University Hospital Tübingen University, Germany, Tübingen, Germany
- Aretaieion University Hospital, Athens, Greece
- Tel Aviv Medical Center, Tel Aviv, Israel
- Spain (2):
  - Hospital Vall d Hebron, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Carson JL, Carless PA, Hebert PC. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2012 Apr 18;4(4):CD002042. doi: 10.1002/14651858.CD002042.pub3. PMID 22513904
- [Background] Corwin HL, Gettinger A, Pearl RG, Fink MP, Levy MM, Abraham E, MacIntyre NR, Shabot MM, Duh MS, Shapiro MJ. The CRIT Study: Anemia and blood transfusion in the critically ill--current clinical practice in the United States. Crit Care Med. 2004 Jan;32(1):39-52. doi: 10.1097/01.CCM.0000104112.34142.79. PMID 14707558
- [Background] Gombotz H, Rehak PH, Shander A, Hofmann A. Blood use in elective surgery: the Austrian benchmark study. Transfusion. 2007 Aug;47(8):1468-80. doi: 10.1111/j.1537-2995.2007.01286.x. PMID 17655591
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Background] Hsieh FY, Bloch DA, Larsen MD. A simple method of sample size calculation for linear and logistic regression. Stat Med. 1998 Jul 30;17(14):1623-34. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-s. PMID 9699234
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Johansson PI, Bochsen L, Stensballe J, Secher NH. Transfusion packages for massively bleeding patients: the effect on clot formation and stability as evaluated by Thrombelastograph (TEG). Transfus Apher Sci. 2008 Aug;39(1):3-8. doi: 10.1016/j.transci.2008.05.012. Epub 2008 Jun 25. PMID 18583193
- [Background] Marik PE, Corwin HL. Efficacy of red blood cell transfusion in the critically ill: a systematic review of the literature. Crit Care Med. 2008 Sep;36(9):2667-74. doi: 10.1097/CCM.0b013e3181844677. PMID 18679112
- [Background] Netzer G, Liu X, Harris AD, Edelman BB, Hess JR, Shanholtz C, Murphy DJ, Terrin ML. Transfusion practice in the intensive care unit: a 10-year analysis. Transfusion. 2010 Oct;50(10):2125-34. doi: 10.1111/j.1537-2995.2010.02721.x. PMID 20553436
- [Background] Phan HH, Wisner DH. Should we increase the ratio of plasma/platelets to red blood cells in massive transfusion: what is the evidence? Vox Sang. 2010 Apr;98(3 Pt 2):395-402. doi: 10.1111/j.1423-0410.2009.01265.x. PMID 20432517
- [Background] Slonim AD, Joseph JG, Turenne WM, Sharangpani A, Luban NL. Blood transfusions in children: a multi-institutional analysis of practices and complications. Transfusion. 2008 Jan;48(1):73-80. doi: 10.1111/j.1537-2995.2007.01484.x. Epub 2007 Sep 24. PMID 17894792
- [Background] Vincent JL, Baron JF, Reinhart K, Gattinoni L, Thijs L, Webb A, Meier-Hellmann A, Nollet G, Peres-Bota D; ABC (Anemia and Blood Transfusion in Critical Care) Investigators. Anemia and blood transfusion in critically ill patients. JAMA. 2002 Sep 25;288(12):1499-507. doi: 10.1001/jama.288.12.1499. PMID 12243637
- [Background] Zink KA, Sambasivan CN, Holcomb JB, Chisholm G, Schreiber MA. A high ratio of plasma and platelets to packed red blood cells in the first 6 hours of massive transfusion improves outcomes in a large multicenter study. Am J Surg. 2009 May;197(5):565-70; discussion 570. doi: 10.1016/j.amjsurg.2008.12.014. PMID 19393349
- [Background] Meier J, Kozek-Langenecker S, Filipescu D, Pitarch JV, Mallett S, Martus P, Matot I. ESA Clinical Trials Network 2012: ETPOS--European Transfusion Practice and Outcome Study. Eur J Anaesthesiol. 2013 May;30(5):199-201. doi: 10.1097/EJA.0b013e32835f0052. No abstract available. PMID 23571430
- [Result] Meier J, Filipescu D, Kozek-Langenecker S, Llau Pitarch J, Mallett S, Martus P, Matot I; ETPOS collaborators. Intraoperative transfusion practices in Europe. Br J Anaesth. 2016 Feb;116(2):255-61. doi: 10.1093/bja/aev456. PMID 26787795